CLINICAL TRIAL: NCT02481908
Title: a New and Non Invasive Method to Calculate STI ( Systolic Time Intervals) Combined to Valsalva Maneuver in Patient With Acute Exacerbation of COPD
Brief Title: STI Combined to Valsalva Maneuver for the Diagnosis of Left Ventricular Dysfunction in COPD Exacerbations
Acronym: STICOPD
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: STI in COPD
Record Dates: First submitted 2015-05-07; First posted 2015-06-25 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Obstructive Chronic Bronchitis With Acute Exacerbation
Keywords: AECOPD; left ventricular dysfunction; valsalva maneuver; systolic time intervals
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: STI measurements at baseline and under Valsalva maneuver — STI measurements at baseline and under Valsalva maneuver

SUMMARY:
The aim of this investigation was to assess the value of Systolic Time Intervals (STIs) as a method of detecting Left Ventricular Dysfunction (LVD) in patients admitted to the emergency department for cute exacerbations of chronic obstructive pulmonary disease (AECOPD) and whether STIs measured under Valsalva manoeuver (VM) could improve the distinction between patients with LVD and those without LVD.

DETAILED DESCRIPTION:
We included patients admitted to the ED for AECOPD. Measurement of STIs included electromechanical activation time (EMAT), left ventricular ejection time and EMAT/LVET ratio. These were performed at baseline and during the first strain phase of the VM using a computerized phono and electrocardiographic method. The diagnosis of LVD was determined on the basis of clinical examination, echocardiography and brain natriuretic peptide. The values of STIs were compared between patients with and without LVD ; their diagnostic performance was assessed using the area under receiver operating characteristic curve (AUC of ROC).

ELIGIBILITY:
Inclusion Criteria:

* Oxygen Saturation (SPO2) <90%,
* Respiratory Rate >25c/min,
* PaCO2 > 6 kPa et pH< 7.35.

Exclusion Criteria:

* Neurological distress and hemodynamic instability
* Confusion, agitation
* pneumothorax
* Non cooperative patients
* Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a prospective study of patients visiting the emergency department of the hospital Fattouma Bourguiba Monastir with decompensated chronic obstructive pulmonary disease COPD
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
diagnosis of left ventricular dysfunction | during the first day admission in emergency department
  Systolic time intervals measured at baseline and under Valsalva maneuver

CONTACTS AND LOCATIONS:
Overall Officials: SEMIR NOUIRA, Pr, Principal Investigator — Fattouma Bourguiba University Hospital
Locations (1):
- CHU Fattouma Bourguiba, Monastir, Tunisia